CLINICAL TRIAL: NCT03040037
Title: Prospective Registry of Atrial Fibrillation Cryoballoon Ablation in the Russian Federation
Brief Title: Cryoballoon Atrial Fibrillation Ablation Registry
Status: Completed | Type: Observational
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Collaborators: RUSSIAN SOCIETY OF CARDIOLOGY (Unknown)
Responsible Party: Sponsor
Other Study IDs: PRAF-CA
Record Dates: First submitted 2016-12-05; First posted 2017-02-01 (Estimated); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
This is a prospective registry of atrial fibrillation cryoablation in the Russian Federation. This study is observational, prospective, multicenter, open-label

DETAILED DESCRIPTION:
The purpose of this Registry is to describe characteristics of patients undergoing cryoballoon ablation, diversity of cryoablation techniques among different centers; to evaluate efficacy and safety of the procedure in the centers with different levels of experience.

ELIGIBILITY:
Inclusion Criteria:

* The indications for catheter ablation of atrial fibrillation
* Signed informed consent to participate in the Register
* Patients undergoing cryoballoon ablation

Exclusion Criteria:

* Left atrial thrombosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult Patient with Indications for Catheter Ablation of Atrial Fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Freedom from arrhythmia: Number of participants with no evidence of atrial achyarrhythmia longer than 30 s, as detected by regular ECG monitoring | 1 Year
  ECG monitoring will be performed in accordance with sites' routine practices (Holter monitoring every 3 months, implantable loop recorder, cardiac rhythm management device interrogation, other regular ECG screening)

SECONDARY OUTCOMES:
Number of participants with adverse events that are related to treatment (i.e. cardiac tamponade, periprocedural stroke, pulmonary vein stenosis, esophageal damage, etc) | 1 Year
Number of participants with adverse events that are related to underlying disease (cardiovascular events not related to atrial fibrillation cryoablation) | 1 Year
Atrial fibrillation procedure characteristics: Mean total ablation procedure time in minutes, mean fluoroscopy time in minutes (during the ablation procedure) | Above parameters will be assessed only during the procedure of cryoablation
  Data will be collected using a web-based system of electronic case report forms
Number of participants with antiarrhythmic drug treatment at 12 months | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution "V. A. Almazov Federal North-West Medical Research Centre" of the Ministry of Health of the Russian Federation, Saint Petersburg, Russia